CLINICAL TRIAL: NCT03581175
Title: IMPlementing Split Regimen OVEr Single Dose
Brief Title: Barriers and Breakthroughs in IMPlementing Split Regimen OVEr Single Dose
Acronym: IMPROVES
Status: Completed | Type: Observational
Sponsor: S. Andrea Hospital (Other)
Responsible Party: Principal Investigator, Emilio Di Giulio, Head of Endoscopy Unit, S. Andrea Hospital
Other Study IDs: 112-2013
Record Dates: First submitted 2018-06-14; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Colonoscopy: Bowel Preparation
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cycle1: Patients undergoing colonoscopy with full bowel cleansing before the improvement phase
  Interventions: Procedure: Colonoscopy; Drug: Bowel cleansing regimen
- Cycle2: Patients undergoing colonoscopy with full bowel cleansing after the improvement phase
  Interventions: Procedure: Colonoscopy; Drug: Bowel cleansing regimen

INTERVENTIONS:
Procedure: Colonoscopy
Drug: Bowel cleansing regimen

SUMMARY:
The split-dose regimen (SpD) has demonstrated its superiority over the day-before regimen (DB) in determining a better colon cleansing and is considered the standard bowel preparation for colonoscopies by the American Society for Gastrointestinal Endoscopy (ASGE) and the European Society of Gastrointestinal Endoscopy (ESGE) guidelines. However its application is still suboptimal due to concerns about patient acceptability, fluid aspiration due to residual gastric contents and challenging viability for early morning colonoscopies. Barriers precluding the prescription of SpD have been explored in few studies mainly in the setting of auditing of current practice, while corrective measure aiming at changing this practice have been prospectively tested in very few, small and selected, cohorts. The present study has the aim of surveying split-dose regimen adoption rate among several endoscopic centres before and after an improvement phase following a plan-do-study-act approach, in order to analyse and correct factors preventing its adoption. A multivariate analysis was planned in order to use collected data to infer factors favouring and limiting split-dose regimen adoption.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing colonoscopy with full bowel cleansing

Exclusion Criteria:

* Incapacity to give informed consent
* Partial colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every inpatient or outpatient undergoing a complete colonoscopy with full bowel cleansing for any indication in one of the participating centres in Central Italy
Sampling Method: Probability Sample
Enrollment: 8267 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Number of participants adopting a split-dose regimen in Cycle1 | 6 months
Number of participants adopting a split-dose regimen in Cycle2 | 3 months
Change from Cycle1 in the proportion of patients adopting a split-dose regimen during Cycle2 after an improvement phase | 9 months (Cycle1 = 6 months + Cycle2 = 3 months, separated by a 21-month improvement phase)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Background] ASGE Standards of Practice Committee; Saltzman JR, Cash BD, Pasha SF, Early DS, Muthusamy VR, Khashab MA, Chathadi KV, Fanelli RD, Chandrasekhara V, Lightdale JR, Fonkalsrud L, Shergill AK, Hwang JH, Decker GA, Jue TL, Sharaf R, Fisher DA, Evans JA, Foley K, Shaukat A, Eloubeidi MA, Faulx AL, Wang A, Acosta RD. Bowel preparation before colonoscopy. Gastrointest Endosc. 2015 Apr;81(4):781-94. doi: 10.1016/j.gie.2014.09.048. Epub 2015 Jan 14. No abstract available. PMID 25595062